CLINICAL TRIAL: NCT01071928
Title: A Phase II Trial of Docetaxel Plus ASA404 as Second-Line Therapy in Patients With Advanced Urothelial Carcinoma: Hoosier Oncology Group GU09-144
Brief Title: Second-Line Docetaxel + ASA404 for Advanced Urothelial Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy of experimental treatment
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Matthew Galsky, Principal Investigator, Hoosier Cancer Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU09-144
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Urothelial Carcinoma
Keywords: Advanced Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Docetaxel; vadimezan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel and ASA404 in Combination (Experimental)
  Interventions: Drug: Docetaxel; Drug: ASA404

INTERVENTIONS:
Drug: Docetaxel — Docetaxel IV 75 mg/m2 over approximately 60 minutes on Day 1
Drug: ASA404 — ASA404 (given after Docetaxel)IV 1800 mg/m2 over approximately 20 minutes on Day 1

SUMMARY:
The purpose of this study is to explore the safety and activity of docetaxel + ASA404 as second-line chemotherapy in patients with advanced urothelial carcinoma.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

21 Day Cycle Treatment Regimen:

* Docetaxel IV 75 mg/m2 over approximately 60 minutes on Day 1
* ASA404 (given after Docetaxel) IV 1800 mg/m2 over approximately 20 minutes on Day 1

Treatment will continue until disease progression or intolerable treatment related adverse effects.

Karnofsky performance status of ≥ 70% within 7 days prior to registration for protocol therapy.

Life Expectancy: Not specified

Hematopoietic:

* Hemoglobin (Hgb) > 9 g/dL
* Platelets > 100 K/mm3
* Absolute neutrophil count (ANC) > 1.5 K/mm3
* INR or Prothrombin Time (PT) < 1.5 x ULN

Hepatic:

* Bilirubin < 1.5 x ULN
* Aspartate aminotransferase (AST, ALT) < 2.5 x ULN

Renal:

* Calculated creatinine clearance of > 45 cc/min using the Cockcroft-Gault formula

Cardiovascular:

* No congestive heart failure (NY Heart Association class III or IV)
* No myocardial infarction within 12 months of study registration for protocol therapy or with implanted cardiac pacemaker
* No unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of transitional cell carcinoma (TCC) of the bladder, urethra, ureter, or renal pelvis (urothelial carcinoma). Histology may be mixed, but still requires a component of TCC.
* Measurable disease according to RECIST (version 1.1) and obtained by imaging within 30 days prior to registration for protocol therapy. Note: Sites of measurable disease can not be within a previously irradiated site.
* Written informed consent and HIPAA authorization for release of personal health information.
* Age > 18 years at the time of consent.
* Must have received only one prior chemotherapy regimen, which must have included one of the following chemotherapeutic agents: cisplatin, carboplatin, or gemcitabine. Note: Prior chemotherapy may have been administered in the perioperative (neoadjuvant/adjuvant) or advanced/metastatic setting. Patients may have received prior treatment with paclitaxel.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 12 weeks after treatment discontinuation.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to registration for protocol therapy.
* Females must not be breastfeeding.

Exclusion Criteria:

* No prior treatment with docetaxel.
* No symptomatic brain metastases. Patients with neurological symptoms must undergo a head CT scan or brain MRI to exclude brain metastasis. NOTE: Patients with treated brain metastasis must be off steroids and have completed radiation at least 14 days prior to registration for protocol therapy.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, Gleason < grade 7 prostate cancers, or other cancers for which the patient has been disease-free for at least 5 years
* No treatment with any investigational agent or chemotherapeutic agent within 30 days prior to registration for protocol therapy.
* No radiotherapy within 14 days prior to registration for protocol therapy. Patients must have recovered from all radiotherapy-related toxicities.
* No major surgery within 30 days prior to registration for protocol therapy (major surgery is defined by the use of general anesthesia).
* No minor surgery 14 days prior to registration for protocol therapy. NOTE: Insertion of a vascular access device is allowed.
* No history of any medical condition resulting in ≥ CTC grade 2 dyspnea.
* Patients without long QT syndrome
* No history of labile hypertension or poor compliance with anti-hypertensive regimen NOTE: No patients with systolic BP >140 mm Hg and/or diastolic BP > 90 mm Hg while on medication for hypertension.
* No presence of atrial tachyarrhythmia (e.g., atrial fibrillation, atrial flutter, multifocal atrial tachycardia, supraventricular tachycardia) if not effectively rate-controlled.
* No history of a sustained ventricular tachycardia
* No history of ventricular fibrillation or Torsades de Pointes
* No right bundle branch block and left anterior or posterior hemiblock (bifascicular block)
* No bradycardia defined as heart rate <50 beats per minute
* No concomitant use of drugs with risk of causing Torsades de Pointes.
* No concomitant use of drugs that are inducers and inhibitors of UGT1A9 and UGT2B7.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine the best overall response rate (as measured by RECIST version 1.1) of docetaxel + ASA404 as second line therapy in patients with advanced urothelial carcinoma. | 12 months

SECONDARY OUTCOMES:
To evaluate progression-free survival in patients with advanced urothelial carcinoma | 12 months
To evaluate survival at 1 year from start of treatment in patients with advanced urothelial carcinoma treated with docetaxel + ASA404 as second line therapy | 12 months
To evaluate the safety of docetaxel and ASA404 combination, as measured by the NCI Common Toxicity Criteria version 3.0 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, M.D., Study Chair — Hoosier Cancer Research Network